CLINICAL TRIAL: NCT01240616
Title: Nicotinic Modulation of the Default Network of Resting Brain Function
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911461; 11-DA-N461
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-12-24

CONDITIONS: Nicotine Dependence
Keywords: Nicotine; Mecamylamine; Attention; fMRI; Default Network; Healthy Volunteer; HV
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- A brain circuit called the default network is the brain circuit that is active when the brain is at rest; that is, when individuals are not concentrating on specific tasks. Previous research has shown that the default network functions differently in people with schizophrenia and Alzheimer s disease, and may contribute to the problems with memory and concentration that can affect people who have these conditions. Studies have also shown that nicotine affects the default network, but more research is needed on the ways in which nicotinic receptors may change activity in these regions and thereby affect individuals ability to concentrate on specific tasks.

Objectives:

- To determine whether and how nicotine and mecamylamine, a drug that blocks nicotinic receptors, affect the default network in nonsmokers in ways that improve thinking and concentration.

Eligibility:

* Healthy, right-handed volunteers between 21 and 50 years of age.
* Volunteers must not have used any kind of tobacco product in the past 2 years.

Design:

* This study involves an initial screening visit, a training visit, and three testing visits.
* Participants will be screened with a medical history and physical examination, as well as blood and urine samples and questions about smoking history.
* Participants will have an initial training session to practice the tasks that will be done during magnetic resonance imaging scans at the testing visits. These tasks will test participants concentration and memory.
* Participants will have three test sessions with the following combinations of study drugs: (1) a nicotine patch and a placebo capsule, (2) a placebo patch and a capsule of mecamylamine, or (3) a placebo patch and capsule. Different combinations will be given at each visit, and participants will not know which one they receive.
* Participants will perform the same concentration and memory tasks at each testing visit, and will provide a blood sample after each visit to determine levels of nicotine and mecamylamine.

DETAILED DESCRIPTION:
Objective: To evaluate the potential of manipulating activity in the so-called default network of resting brain function by nicotinic ligands. Default network activity modulates cognitive functioning, and effects of nicotine thereon may motivate smoking behavior. In the future, this mechanism could become a novel approach to improving cognition in disease populations that show dysfunction of this network, such as schizophrenia or Alzheimer s disease.

Study population: 27 healthy non-smokers.

Design: A double-blind, placebo-controlled, within-subject fMRI study, evaluating regional brain activation and cognitive functions under conditions of transdermal nicotine (7 mg/day), oral mecamylamine (a nicotinic antagonist, 7.5 mg), and placebo.

Outcome measures: Activity and functional connectivity of default regions during cognitive task performance, measures of cognitive task performance, measures of subjective state, and plasma concentrations of nicotine, nicotine metabolites and mecamylamine.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 21 through 55. We want to avoid exposing a maturing brain to centrally active substances that it has not previously been exposed to (non-smokers), and to increase sensitivity for measuring drug effects by minimizing population inhomogeneity related to both cognitive decline with normal aging (Verhaeghen and Salthouse 1997, De Luca et al. 2003) and to ongoing brain maturation.
  2. Did not consume cigarettes, cigarillos, cigars, or other tobacco or nicotine-containing products more than 20 times in lifetime, and did not use any nicotine-containing product at all within the last two years.
  3. Normal or corrected to normal vision (at least 20/80).

EXCLUSION CRITERIA:

1. Presence of metal objects in the body, implanted electronic devices, or any other counter indication for MRI.
2. Claustrophobia.
3. Major psychiatric disorders including mood, anxiety or psychotic disorders.
4. Cardiovascular or cerebrovascular disease, such as history of myocardial infarction, heart failure, angina, stroke, severe arrhythmias, or EKG abnormalities as specified under Screening methods .
5. Kidney or liver disease.
6. Hypertension (resting systolic BP above 140 or diastolic above 85 mm Hg).
7. Hypotension (resting systolic BP below 95 or diastolic below 60).
8. Use of any prescription or over-the-counter drug other than supplements and birth control.
9. History of or current neurological illnesses, such as stroke, seizures, dementia or organic brain syndrome.
10. Learning disability, attention deficit disorder, or any other condition that impedes memory and attention.
11. Glaucoma, organic pyloric stenosis, uremia or renal insufficiency (see Mecamylamine-related risks).
12. Prostatic hypertrophy, bladder neck obstruction or urethral stricture (see Mecamylamine-related risks).
13. Left-handed or ambidextrous.
14. Pregnant as determined by urine test, or breast-feeding.
15. History or current diagnosis of drug or alcohol abuse or dependence.
16. IQ < 85 as estimated by the WASI vocabulary subtest.
17. Strong disposition to get car sick.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2010-10-24; Study Completion 2014-12-24

PRIMARY OUTCOMES:
Activity and functional connectivity of default regions during cognitive task performance, measures of cognitive task performance, measures of subjective state, and plasma concentrations of nicotine, nicotine metabolites and mecamylamine.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland
  - University of Maryland at Baltimore/MPRC, Catonsville, Maryland

REFERENCES:
- [Background] Binder JR, Frost JA, Hammeke TA, Bellgowan PS, Rao SM, Cox RW. Conceptual processing during the conscious resting state. A functional MRI study. J Cogn Neurosci. 1999 Jan;11(1):80-95. doi: 10.1162/089892999563265. PMID 9950716
- [Background] Bluhm RL, Miller J, Lanius RA, Osuch EA, Boksman K, Neufeld RW, Theberge J, Schaefer B, Williamson P. Spontaneous low-frequency fluctuations in the BOLD signal in schizophrenic patients: anomalies in the default network. Schizophr Bull. 2007 Jul;33(4):1004-12. doi: 10.1093/schbul/sbm052. Epub 2007 Jun 7. PMID 17556752
- [Background] Boyajian RA, Otis SM. Acute effects of smoking on human cerebral blood flow: a transcranial Doppler ultrasonography study. J Neuroimaging. 2000 Oct;10(4):204-8. doi: 10.1111/jon2000104204. PMID 11147398